CLINICAL TRIAL: NCT02453074
Title: Automated System for Gathering and Reporting Clinical Outcomes to Providers
Status: Completed | Type: Observational
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Ben Gross, Ben Gross, Harvard Medical School (HMS and HSDM)
Other Study IDs: 2014P002351
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Ambulatory Care

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Online survey - Follow up for Better Care

SUMMARY:
The purpose of this study is to design and test the feasibility of a system to survey patients regarding the outcome of acute care visits and to report back to the healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older visiting participating primary care clinics who agree to be contacted by email to complete a survey on clinical outcomes.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of two primary clinics at Massachusetts General Hospital, Boston MA
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Survey response rate | Assessed at the end of the 12 week study period